CLINICAL TRIAL: NCT01277289
Title: Multicenter, Randomized, Double-blind, Parallel-group Study of Intra-erythrocyte Dexamethasone Versus Placebo in Patients With Steroid-dependent Crohn's Disease
Brief Title: Intra-erythrocyte Dexamethasone Versus Placebo in Patients With Steroid-dependent Crohn's Disease
Acronym: Crodex
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: due to the difficulty to enroll suitable patients
Sponsor: Quince Therapeutics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Crodex01; 2008-007329-38 (EudraCT Number)
Record Dates: First submitted 2011-01-05; First posted 2011-01-14 (Estimated); Results first posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2023-12

CONDITIONS: Crohn's Disease
Keywords: dexamethasone; ery-dex; Chron's disease; CD
MeSH Terms: conditions — Crohn Disease | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ery-dex (Experimental): Ery-dex (dexamethasone sodium phosphate)is administered as intra-erythrocyte drug at monthly interval
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): placebo comparator (sodium chloride instead of dexamethasone sodium phosphate) is administered in infusion at monthly interval.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — 500 mg/20 ml encapsulated in erythrocytes, every month for 12 months
  Other Names: Ery-dex

SUMMARY:
Primary objective:

Assessment of the efficacy of EryDex vs PLACEBO in maintaining patients with steroid-dependent Crohn's disease in clinical remission throughout 12 months without oral steroids.

Secondary objectives:

1. safety of EryDex
2. emergence of new adverse effects from steroids or disappearance of those possibly pre-existing in the various subgroups of patients;
3. duration of the period of remission;
4. evaluation of the hypophysis-adrenal function;
5. study of plasma concentrations of dexamethasone;
6. effect of therapy on the metabolism of calcium and on indexes of inflammation;
7. assessing the quality of life;
8. rate of surgical resection
9. evaluation of the indirect costs of care.

DETAILED DESCRIPTION:
This was a multicenter, randomized, double-blind, PLACEBO-controlled, parallel-group study comparing EryDex versus PLACEBO. Patients with steroid-dependent Crohn's disease were enrolled and randomized to undergo 12 infusions of intraerythrocyte dexamethasone (EryDex), or PLACEBO. A balanced (1:1) randomization between the two treatment groups (EryDex / PLACEBO) was employed.

At the time of randomization, study patients were stratified at each study site according to their previous therapy with AZT/6MP/MTX (never treated with AZT/6MP/MTX or intolerant/resistant to the therapy with AZT/6MP/MTX). The treatment was planned to be performed with 12 monthly infusions of EryDex or PLACEBO.

Patients were followed-up after completion of the treatment for 6 months in patients regularly completing the study and 3 months in patients discontinuing from the study prematurely. The evaluation of the primary and secondary objectives was to be done at the 12th month of study (one month after the last study drug infusion), or upon relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects;
2. Age > 18 years;
3. Patients with steroid-dependent Crohn's disease, documented in the medical history, having suffered from at least one episode of relapse (CDAI > 150) in the last 12 months. Patients should have been in clinical remission (CDAI < 150) for at least four weeks, on stable therapy with at least 10 mg of methylprednisolone (or equivalent), or been on steroidal tapering after a recent relapse. Patients with intolerance or resistance to AZT/6-MP/MTX were eligible;
4. Patients willing and able to give written informed consent.

Exclusion Criteria:

1. Patients with Crohn's disease with intestinal sub-occlusion, or suspect of abdominal abscess, or with active perianal disease, or with clinically active disease at randomization (CDAI ≥150);
2. Patients already on therapy with immunosuppressant agents (AZT, 6-MP, MTX) for less than 4 months;
3. Patients having received therapy with infliximab (or other anti-TNF) in the previous 3 months;
4. Investigational treatments in the previous 3 months prior to randomization;
5. Pregnant women, or women who were not using valid birth-control measures, except those in surgical menopause; breast feeding;
6. Non collaborating subjects or those unable to be compliant with the treatment and the study schedules;
7. Severe concomitant diseases such as :

   1. patients with inadequate "bone marrow reserve": WBC < 3000 /mm3; PLTs < 75000 /mm3; Hb < 8 g/dl
   2. liver disease with total bilirubin ≥ 3 times the upper limit of normal (ULN), AST (GOT) ≥ 3x ULN, alkaline phosphatase ≥ 3x ULN
   3. renal disease with serum creatinine ≥ 3 mg/dl
   4. serious cardiac, allergic, lung, neurological diseases, neoplastic or pre-neoplastic disease
   5. diseases (other than Crohn's) requiring chronic steroid treatment;
8. Elective surgery already scheduled at the start of the study (NB: patients having undergone previous surgery for Crohn's disease could be enrolled, if the patient had fully recovered and had been in remission for at least 4 weeks);
9. Chronic use of alcohol; drug addiction;
10. Subjects with contra-indication to the use of steroids (i.e. systemic fungal infections);
11. Evidence of clostridium difficilis in the stools.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-06-03 (Actual); Primary Completion 2011-12-30 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Andriulli, MD, Principal Investigator — Unafilliated
Locations (8):
- Italy (6):
  - Policlinico Sant'Orsola, Bologna
  - Ospedale Careggi, Florence
  - Ospedale Cervello, Palermo
  - Complesso Integrato Columbus, Rome
  - Ospedale San Camillo, Rome
  - A.O. San Donato, San Donato Milanese
- Spitalul Clinic Judetean De Urgenta, Cluj-Napoca, Romania
- Clinic CIBER EHD, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 63 patients enrolled into the screening phase at 10 sites; of these, 51 patients (representing the Safety population) were randomized at 9 sites.
Period: Overall Study
Arm/Group | Ery-dex | Placebo
Started | 28 | 23
Completed | 5 | 2
Not Completed | 23 | 21
Not completed — fragile vein | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — therapy failure and/or Crohn's surgery | 13 | 16
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 2 | 1
Not completed — consent withdrawn | 1 | 1
Not completed — premature closure of the study | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ery-dex | Placebo | Total
Number analyzed (Participants) | 28 | 23 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 20 | 44
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (14.9) | 43.4 (12.5) | 45.5 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 7 | 27
  Male | 8 | 16 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 23 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Romania | 1 | 0 | 1
  Italy | 27 | 22 | 49
  Spain | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Maintaining Steroids-free Clinical Remission (CDAI<150) Without Surgery for 12 Months
Description: Clinical remission was defined as a Crohn's Disease Activity Index (CDAI) < 150. A therapy failure was considered to have occurred in patients with a CDAI score over 150 for > 2 weeks and/or the need for systemic steroids (with / without surgery). Hence, the higher the index, the worse the outcome.
Time Frame: after 12 months
Population: Safety population, defined as all randomized patients who took at least one dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Ery-dex | Placebo
Number analyzed (Participants) | 28 | 23
Participants | 5 | 2

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: This evaluation of safety was made by the comparison of treatment emergent adverse events (TEAE). Treatment emergent adverse events (TEAE) are undesirable events not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment.
Time Frame: after 12 months
Population: Safety population, defined as all randomized patients who took at least one dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Ery-dex | Placebo
Number analyzed (Participants) | 28 | 23
Participants | 13 | 6

3. Secondary Outcome: Percentage of Patients Interrupting the Study Because of Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: after 12 months
Population: Safety population, defined as all randomized patients who took at least one dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Ery-dex | Placebo
Number analyzed (Participants) | 28 | 23
Participants | 2 | 1

4. Secondary Outcome: Duration of the Period of Steroid-free Clinical Remission
Description: The mean time between the end of the steroid therapy and a confirmed relapse of the disease.
Time Frame: From end of the steroid therapy to relapse, up to 545 days
Population: Data reported only for 9 subjects for the EryDex group and for 13 subjects in the placebo group of the safety set. For the remaining subjects, data are not included because of no treatment with steroids, or no last date available on the use of steroids, or steroids still ongoing.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ery-dex | Placebo
Number analyzed (Participants) | 9 | 13
Days | 55.3 (73.2) | 84.9 (72.9)

5. Secondary Outcome: Dosing of Serum Cortisol
Description: Levels of serum cortisol were measured at baseline and following Adrenocorticotropic Hormone (ACTH) trigger.
Time Frame: At Baseline and at the end of the study (18 months)
Population: Safety Set defined as all randomized patients who took at least one dose of the study medication
Measure: Mean (Standard Deviation); unit: μg/dl
Arm/Group | Ery-dex | Placebo
Number analyzed (Participants) | 28 | 23
μg/dl
  At Baseline - before ACTH | 6.8 (4.6) | 7.1 (6.2)
  At the end of the study - before ACTH | 11.3 (8.6) | 6.4 (5.4)
  At baseline - after ACTH | 10.3 (7.6) | 11.0 (6.5)
  At the end of the study - after ACTH | 18.4 (4.7) | 12.7 (7.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Visit 1 ( Day 15) up to Visit 15 (Day 600)
Description: TEAEs were defined as those events with an onset any time following the first dose of trial medication up to 30 days after last dose of trial medication or those starting before the treatment period but continuing and worsening during the treatment period or leading to treatment discontinuation (even if temporary).
Arm/Group | Ery-dex | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 1/23
Serious Adverse Events (participants affected / at risk) | 6/28 | 4/23
Other Adverse Events (participants affected / at risk) | 19/28 | 16/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ery-dex (N=28) | Placebo (N=23)
Crohn's disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 3 (3)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ery-dex (N=28) | Placebo (N=23)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Cushingoid (Endocrine disorders) | 4 (4) | 0 (0)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1)
Acetonaemic vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Anal Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (7)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Rectal tenesmus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 2 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Asthenia (General disorders) | 3 (4) | 4 (5)
Hyperpyrexia (General disorders) | 2 (3) | 0 (0)
Irritability (General disorders) | 3 (3) | 2 (2)
Oedema (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster ophthalmic (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood iron decreased (Investigations) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (10)
Affect lability (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Influenza (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (5)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin striae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No